CLINICAL TRIAL: NCT03168802
Title: Comparative Study of Magnetic Resonance-guided Focused Ultrasound and Radiofrequency Ablation for Treatment of Facet-joint Osteoarthritis Low Back Pain
Brief Title: MRgFUS and RFA for Treatment of Facet-joint Osteoarthritis Low Back Pain
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Taipei Medical University Hospital (Other)
Responsible Party: Principal Investigator, Meng-Huang Wu, Principal Investigator, Taipei Medical University Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: N201609021
Record Dates: First submitted 2017-04-10; First posted 2017-05-30 (Actual); Last update posted 2024-12-05 (Actual); Status verified 2024-12

CONDITIONS: Chronic Low Back Pain; Facet Joint Syndrome
Keywords: Focused ultrasound Ablation; Radiofrequency Ablation; Facet joint syndrome; Chronic low back pain
MeSH Terms: interventions — Radiofrequency Ablation

STUDY DESIGN:
Intervention Model Description: 50 patients in each arm.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- MRgFUS facet treatment (Experimental): MRgFUS ablation for facet joint pain once at Lumbar spine
  Interventions: Procedure: MRgFUS ablation
- Radiofrequency ablation facet treatment (Active Comparator): Radiofrequency ablation for facet joint pain once at Lumbar spine
  Interventions: Procedure: Radiofrequency ablation

INTERVENTIONS:
Procedure: MRgFUS ablation — Focus ultrasound ablation therapy under MRI navigation for facet joint syndrome.
  Arms: MRgFUS facet treatment
Procedure: Radiofrequency ablation — Radiofrequency ablation therapy under C-arm navigation for facet joint syndrome.
  Arms: Radiofrequency ablation facet treatment

SUMMARY:
This is a prospective, randomized, two-arm, phase II study.

The purpose of this study is:

* To evaluate and compare the efficacy and safety of magnetic resonance-guided focused ultrasound (MRgFUS) and radiofrequency ablation (RFA) for treatment of facet-joint osteoarthritis low back pain.
* Determining the effect of the MRgFUS System and RFA for improving functional disabilities and in reducing pain resulting from facet-joint osteoarthritis low back pain. Efficacy will be determined by the level of pain relief (as measured by the Numerical Rating Scale, NRS), decrease in analgesics/opiate, improved quality of life (as measured by the Oswestry Disability Questionnaire, ODQ, and core outcome measures index questionnaire, COMI), pain interference with function (as measured by the Brief Pain Inventory-Interference scale, BPI-QoL), general health status (as measured by the EQ5D), physical exam, X-ray and MRI studies from baseline up to 12-Months post- MRgFUS and radiofrequency treatment.
* Evaluate incidence and severity of adverse events associated with the MRgFUS system and RFA used for the treatment of pain resulting from facet-joint osteoarthritis low back pain.

ELIGIBILITY:
Inclusion Criteria:

1. Men and women age 20 to 79 years old
2. Suffering from lumbar vertebral facet joint syndrome.
3. Lower back pain at least six months (NRS≥4).
4. Conventional treatment of pain includes NSAIDs, opioids, muscle relaxants, oral steroids, physical therapy or chiropractic therapy.
5. Imaging of the spine have facet osteoarthritis.
6. Referred pain is no more below the knee.
7. At least once when local anesthesia or diagnostic medial nerve branch injection, pain reduction> 75% (0.5ml of 2% lidocaine).

Exclusion Criteria:

1. Patients with evidence of lumbosacral radiculopathy on MRI, CT or physical exam findings, including radicular leg pain.
2. Patients with motor deficit or any other indication for surgical intervention.
3. Patients with MRgFUS or RF treatment for LBP within the last 6 months.
4. Patients with previous low back surgery.
5. Patients who are pregnant.
6. Patients with existing malignancy.
7. Patients with allergies to relevant contrast, anesthetics, sedation drugs.
8. Patients with contraindications for MRI.
9. Patients with an acute medical condition (e.g., pneumonia, sepsis) that is expected to hinder them from completing this study.
10. Patients with unstable cardiac status including:

    * Unstable angina pectoris on medication
    * Patients with documented myocardial infarction less than 40 days prior to protocol enrolment
    * Patients with Severe Congestive Heart Failure, NYHA class 4.
    * Patients on anti-arrhythmic drugs or with uncontrolled and/or untreated arrhythmia status
    * Patients with pacemaker
11. Patients with severe cerebrovascular disease (CVA within last 6 months)
12. Patients with severe hypertension (diastolic BP > 100 on medication)
13. Patients with an active infection or severe hematological, neurological, or other uncontrolled disease.
14. Patients unable to communicate with the investigator and staff.
15. Patients who are not able or willing to tolerate the required prolonged stationary position during treatment (approximately 2 hrs.)
16. Coagulation disorders or other bleeding disorders, use of anticoagulants or antiplatelet drugs within 5 days before treatment.
17. When local anesthesia or diagnostic medial nerve branch injection, the pain does not reach 75% (0.5 mL of 2% lidocaine).

Ages: 20 Years to 79 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2018-08-24 (Actual); Primary Completion 2025-11-25 (Estimated); Study Completion 2025-11-25 (Estimated)

PRIMARY OUTCOMES:
Pain score change: Numerical Rating Scale (NRS) | 24-week post-treatment
  Efficacy

SECONDARY OUTCOMES:
Pain score change: Numerical Rating Scale (NRS) | 1-, 4-, 8-, 12-, 36-, 52-week post-treatment
  Efficacy
Functional scales change: Brief Pain Inventory-Quality of Life (BPI-QoL) | 1-, 4-, 8-, 12-, 24-, 36-, 52-week post-treatment
  Efficacy
Functional scales change: Oswestry Disability Questionnaire (ODQ) | 1-, 4-, 8-, 12-, 24-, 36-, 52-week post-treatment
  Efficacy
Functional scales change: Core Outcome Measurement Index (COMI) | 1-, 4-, 8-, 12-, 24-, 36-, 52-week post-treatment
  Efficacy
Functional scales change: EQ5D Quality of Life questionnaires | 1-, 4-, 8-, 12-, 24-, 36-, 52-week post-treatment
  Efficacy
Amount of analgesic consumption | 1-, 4-, 8-, 12-, 24-, 36-, 52-week post-treatment
  Efficacy
Adverse event | 1-, 4-, 8-, 12-, 24-, 36-, 52-week post-treatment
  Safety

OTHER OUTCOMES:
Physical exams for back range of motion | 1-, 4-, 8-, 12-, 24-, 36-, 52-week post-treatment
  Efficacy
X-ray for spine facet change | 1-, 4-, 8-, 12-, 24-, 36-, 52-week post-treatment
  Efficacy

CONTACTS AND LOCATIONS:
Overall Officials: Yen Yun, PhD, Study Chair — Taipei Medical University
Locations (1):
- Taipei medical university hospital, Taipei, Please Select, Taiwan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Weeks EM, Platt MW, Gedroyc W. MRI-guided focused ultrasound (MRgFUS) to treat facet joint osteoarthritis low back pain--case series of an innovative new technique. Eur Radiol. 2012 Dec;22(12):2822-35. doi: 10.1007/s00330-012-2628-6. Epub 2012 Aug 31. PMID 22935902
- [Background] Kaye EA, Monette S, Srimathveeravalli G, Maybody M, Solomon SB, Gulati A. MRI-guided focused ultrasound ablation of lumbar medial branch nerve: Feasibility and safety study in a swine model. Int J Hyperthermia. 2016 Nov;32(7):786-94. doi: 10.1080/02656736.2016.1197972. Epub 2016 Jul 21. PMID 27443328
- [Background] Krug R, Do L, Rieke V, Wilson MW, Saeed M. Evaluation of MRI protocols for the assessment of lumbar facet joints after MR-guided focused ultrasound treatment. J Ther Ultrasound. 2016 Apr 6;4:14. doi: 10.1186/s40349-016-0057-8. eCollection 2016. PMID 27054038
- [Background] Maas ET, Ostelo RW, Niemisto L, Jousimaa J, Hurri H, Malmivaara A, van Tulder MW. Radiofrequency denervation for chronic low back pain. Cochrane Database Syst Rev. 2015 Oct 23;2015(10):CD008572. doi: 10.1002/14651858.CD008572.pub2. PMID 26495910